CLINICAL TRIAL: NCT06878378
Title: Identification of Risk Factors for Inadequate Bowel Preparation Before Colonoscopy and Construction of a Predictive Model: a Nationwide Multicenter Prospective Study
Brief Title: Risk Factors for Inadequate Bowel Preparation Before Colonoscopy
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Other Study IDs: CHEC2025-083
Record Dates: First submitted 2025-03-13; First posted 2025-03-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colonoscopy; Colonoscopy: Bowel Preparation
Keywords: bowel preparation; colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- outpatients and inpatients scheduled for colonoscopy or polypectomy: The target population includes outpatients and inpatients scheduled for colonoscopy or polypectomy in the gastroenterology departments of participating centers between February 2025 and December 2026. Data from these individuals will be collected to assess factors influencing bowel preparation quality.
  Interventions: Other: Investigation of Factors Influencing Bowel Preparation Quality

INTERVENTIONS:
Other: Investigation of Factors Influencing Bowel Preparation Quality — Observed parameters include BMI, history of abdominal surgery, history of diabetes, history of diarrhea and constipation, stool characteristics, and specific bowel preparation protocols.

SUMMARY:
The primary objectives of this study are twofold:

Firstly, to investigate the current status of bowel preparation protocols and their quality across hospitals at various levels in China, particularly following the release of the updated 2023 bowel preparation guidelines. This aims to standardize and optimize bowel preparation protocols nationwide.

Secondly, to identify and analyze risk factors contributing to suboptimal bowel preparation quality in patients undergoing colonoscopy. The study will examine the correlation between these factors and bowel preparation scores, establish a risk prediction model for preparation failure, and provide a theoretical foundation for developing personalized bowel preparation regimens tailored to individual patient characteristics.

DETAILED DESCRIPTION:
The project is divided into three key phases:

1. Initiation Phase:

   Develop a Bowel Preparation Assessment Questionnaire (BPAQ) to standardize data collection.

   Establish collaborative centers (multicenter hospitals) nationwide for coordinated implementation.
2. Implementation Phase:

   Conduct on-site audits to evaluate bowel preparation practices across participating centers.

   Deliver protocol-specific training to healthcare providers, emphasizing compliance with the 2023 guidelines.

   Systematically collect bowel preparation data, including patient demographics, protocol adherence metrics, and clinical outcomes.
3. Conclusion Phase:

Prioritize data quality assurance through dual-entry validation and logic checks to ensure authenticity, comprehensiveness, and objectivity.

Generate consolidated reports to identify systemic gaps and propose evidence-based optimization strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years, regardless of gender, scheduled for colonoscopy
* Written informed consent has been obtained

Exclusion Criteria:

* History of acute myocardial infarction (within 6 months), severe cardiac/hepatic/renal insufficiency, or psychiatric disorders
* Current use of anticoagulants (e.g., aspirin, warfarin) or presence of coagulation disorders
* Pregnancy or lactation;
* History of inflammatory bowel disease or acute intestinal infection within the past 2 weeks;
* History of colorectal cancer, familial adenomatous polyposis (FAP), or Peutz-Jeghers syndrome;
* History of intestinal obstruction, perforation, stricture, or other conditions precluding completion of colonoscopy;
* Non-compliance with bowel preparation protocols (e.g., ingestion of <80% of prescribed polyethylene glycol (PEG) electrolyte solution);
* Severe hearing impairment, cognitive dysfunction, or inability to cooperate with the study;
* Prior enrollment in this study with a repeat colonoscopy appointment;
* Current participation in other clinical trials or participation in any trial within the preceding 60 days;
* Refusal to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population includes outpatients and inpatients scheduled for colonoscopy or polypectomy in the gastroenterology departments of participating centers between February 2025 and February 2026.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
adequate bowel preparation rate | The adequate bowel preparation rate can be assessed immediately upon completion of colonoscopy

SECONDARY OUTCOMES:
adenoma detection rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China